CLINICAL TRIAL: NCT06642467
Title: BGEM Use as Blood Glucose Prediction Model in T2DM Population of Indonesia
Status: Completed | Type: Observational
Sponsor: Krida Wacana Christian University (Other)
Collaborators: Actxa (Unknown); Lif (Unknown)
Responsible Party: Sponsor
Other Study IDs: KridaWacanaCU
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Group: Subjects age 18-59 years old who was diagnosed with type 2 diabetes mellitus, or pre DM or known to have abnormal Hba1c or blood glucose results
  Interventions: Device: BGEM
- Non diabetic Group: Subjects age 18-59 years old who never diagnosed to have diabetes mellitus or pre DM
  Interventions: Device: BGEM

INTERVENTIONS:
Device: BGEM — BGEM is an ai driven model to predict blood glucose using ppg sensor

SUMMARY:
Using signals from consumer-grade PPG sensors on wrist wearables, smart rings or hearables, BGEM® AI model computes the relevant digital biomarkers correlated with the change of blood glucose level to predict a blood glucose result for monitoring and evaluating diabetic risks Ukrida in collaboration with Actxa & Lif aims to enhance the current model's prediction accuracy to predict the blood glucose levels of individuals almost as accurately as a glucometer. To achieve this, Actxa aims to collect data from around 500 individuals with diabetes in this exercise and 400 healthy or undiagnosed (prediabetes/diabetes) individuals.

DETAILED DESCRIPTION:
Background Powered by our AI-driven algorithm, the Actxa's Blood Glucose Evaluation and Monitoring (BGEM®) is a cloud-based technology that enables wearables with photoplethysmography (PPG) sensors to monitor and evaluate diabetic risk of individuals regularly in a non-invasive way.

Using signals from consumer-grade PPG sensors on wrist wearables, smart rings or hearables, BGEM® AI model computes the relevant digital biomarkers correlated with the change of blood glucose level to predict a blood glucose result for monitoring and evaluating diabetic risks. Our previous study has shown the potential of using PPG sensors to detect elevated blood glucose levels among a non-diabetic population1.

Objective Ukrida in collaboration with Actxa & Lif to enhance the current model's prediction accuracy to predict the blood glucose levels of individuals almost as accurately as a glucometer. To achieve this, Actxa aims to collect data from around 500 individuals with diabetes in this exercise and 400 healthy or undiagnosed (prediabetes/diabetes) individuals, as part of Actxa's collaboration with UKRIDA Hospital.

With the data collected, our algorithm holds the potential to significantly improve the management of blood glucose levels for people with and without diabetes, ultimately enhancing their overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-59 yo
* diabetic or non diabetic
* healthy enough to undergoes normal daily activity

Exclusion Criteria:

* o Wears a pacemaker

  * Is currently pregnant
  * Has an infection
  * Has a fever

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 500 people of diabetic subjects and 400 people of non diabetic subjects
Sampling Method: Non-Probability Sample
Enrollment: 885 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Prediction value of BGEM | July-December 2024
  Result of predictive model will be compared with blood glucose analysis
Prediction value of BGEM | July-December 2024
  Result of predictive model will be compared with Hba1c

SECONDARY OUTCOMES:
Variables influencing BGEM | July-December 2024
  Analysis to determine any variables from subjects that influence BGEM

CONTACTS AND LOCATIONS:
Locations (1):
- Ukrida Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No